CLINICAL TRIAL: NCT03138811
Title: A Randomized, Subject- and Investigator-blinded, Placebo-controlled, Paralleldesign, Bronchoprovocation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Doses of Inhaled CSJ117 in Adult Subjects With Mild Atopic Asthma
Brief Title: A Bronchoprovocation Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CSJ117 in Adult Subjects With Mild Atopic Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCSJ117X2201; 2016-004929-16 (EudraCT Number)
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Asthma
Keywords: asthma; allergen bronchoprovocation; pharmacodynamics; pharmacokinetics; safety; tolerability
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSJ117 (Experimental): low dose, medium dose, or high dose administered as a once daily inhaled dose
  Interventions: Drug: CSJ117
- Placebo (Placebo Comparator): placebo comparator administered as once daily inhaled dose
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: CSJ117 — inhaled once daily dose
  Arms: CSJ117
Drug: Placebo Comparator — inhaled once daily dose
  Arms: Placebo

SUMMARY:
This is a non-confirmatory, randomized, subject and investigator blinded, placebo-controlled, parallel-design, multi-center bronchoprovocation study. Approximately 55 subjects with mild stable atopic asthma who exhibit an EAR and LAR to a common inhaled allergen will receive multiple once daily doses of inhaled CSJ117 or placebo over 12 weeks. Two sequential dose cohorts are planned for this study, Cohort 1 and Cohort 2. Cohort 2 will be split into two parts, Cohort 2a and 2b

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stable mild atopic asthma, as defined by the American Thoracic Society/ European Respiratory Society statement, who exhibit an early and late asthmatic response to a common inhaled allergen during the screening allergen inhalation challenge.
* Throughout the screening period and at baseline, only infrequent use of inhaled short-acting beta2-agonists (less than or equal to twice weekly) to treat asthma and/or prophylactic use prior to exercise. Inhaled short-acting beta2-agonist must be withheld for 8 hours before spirometry.

Exclusion Criteria:

* Hospitalization or emergency room treatment for acute asthma in the 6 months prior to screening or during the screening period.
* Any worsening or exacerbation of asthma (e.g., an event requiring a change in treatment) in the six weeks before screening or during the screening period.
* A history of any clinically significant chronic pulmonary disease other than mild atopic asthma, including but not limited to COPD, interstitial lung disease or bronchiectasis
* Use of immunosuppressive medications or allergen-specific immunotherapy within 6 months prior to screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Number of adverse events and serious adverse events | 12 weeks
  An AE is the appearance or worsening of any undesirable sign, symptom, or medical condition occurring after starting the study drug even if the event is not considered to be related to study drug. Study drug includes the investigational drug under evaluation and the comparator drug or placebo that is given during any phase of the study. Adverse events starting on or after the time of the first inhalation of study drug are classified as a treatment emergent adverse event.
Late asthmatic response as measured by the AUC for time adjusted percent decrease in FEV1 | 12 weeks
  Late asthmatic response (LAR) is considered a ≥ 15% fall in FEV1 between 3 and 7 hours after an allergen inhalation challenge. The AUC for time adjusted percent decrease in FEV1 will be compared between CSJ117 and placebo groups.
Late asthmatic response as measured by the maximum percentage decrease in FEV1 | 12 weeks
  Late asthmatic response (LAR) is considered a ≥ 15% fall in FEV1 between 3 and 7 hours after an allergen inhalation challenge. The maximum percentage decrease in FEV1 will be compared between CSJ117 and placebo groups.

SECONDARY OUTCOMES:
Early asthmatic response as measured by the time adjusted AUC percent decrease in FEV1 | 6 weeks and 12 weeks
  Early asthmatic response (EAR) is considered a ≥ 20% fall in FEV1 within the 2 hours after an allergen inhalation challenge. The time adjusted AUC percent decrease will be compared between CSJ117 and placebo groups.
Early asthmatic response as measured by the maximum percentage decrease in FEV1 | 6 weeks and 12 weeks
  Early asthmatic response (EAR) is considered a ≥ 20% fall in FEV1 within the 2 hours after an allergen inhalation challenge. The maximum percentage decrease will be compared between CSJ117 and placebo groups.
Early asthmatic response as measured by the minimum of the absolute in FEV1 | 6 weeks and 12 weeks
  Early asthmatic response (EAR) is considered a ≥ 20% fall in FEV1 within the 2 hours after an allergen inhalation challenge. The minimum of the absolute in FEV1 will be compared between CSJ117 and placebo groups.
Late asthmatic response as measured by the time adjusted AUC in FEV1 | 6 weeks
  Late asthmatic response (LAR) is considered a ≥ 15% fall in FEV1 between 3 and 7 hours after an allergen inhalation challenge. The time adjusted in FEV1 will be compared between CSJ117 and placebo groups.
Late asthmatic response as measured by the maximum percentage decrease in FEV1 | 6 weeks
  Late asthmatic response (LAR) is considered a ≥ 15% fall in FEV1 between 3 and 7 hours after an allergen inhalation challenge. The maximum percentage decrease in FEV1 will be compared between CSJ117 and placebo groups.
Late asthmatic response as measured by the minimum absolute FEV1 | 6 weeks and 12 weeks
  Late asthmatic response (LAR) is considered a ≥ 15% fall in FEV1 between 3 and 7 hours after an allergen inhalation challenge. The minimum absolute in FEV1 will be compared between CSJ117 and placebo groups.
Measurement of CSJ117 serum concentration and calculation of Tmax | 12 weeks
  Tmax is the time to reach the maximum concentration after drug administration
Measurement of CSJ117 serum concentration and calculation of Cmax | 12 weeks
  Cmax is the observed maximum plasma concentration following drug administration
Measurement of CSJ117 serum concentration and calculation of AUCtau | 12 weeks
  The area under the plasma (or serum or blood) concentration-time curve from time zero to the end of the dosing interval tau [mass x time / volume]
Measurement of CSJ117 serum concentration and calculation of Ctrough) | 12 weeks
  Ctrough is the observed serum (or plasma or blood) concentration that is just prior to the beginning of, or at the end of, a dosing interval.
Measurement of CSJ117 serum concentration and calculation of Racc | 12 weeks
  Racc is the accumulation ratio
Measurement of CSJ117 serum concentration and calculation of Lambda_z | 12 weeks
  Lambda_z is the apparent elimination rate constant
Measurement of CSJ117 serum concentration and calculation of T1/2 | 12 weeks
  T1/2 is the terminal elimination half-life [time]

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Canada (6):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Saskatchewan, Saskatchewan
  - Novartis Investigative Site, Vancouver
- Germany (4):
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Großhansdorf
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Mainz

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Gauvreau GM, Hohlfeld JM, FitzGerald JM, Boulet LP, Cockcroft DW, Davis BE, Korn S, Kornmann O, Leigh R, Mayers I, Watz H, Grant SS, Jain M, Cabanski M, Pertel PE, Jones I, Lecot JR, Cao H, O'Byrne PM. Inhaled anti-TSLP antibody fragment, ecleralimab, blocks responses to allergen in mild asthma. Eur Respir J. 2023 Mar 9;61(3):2201193. doi: 10.1183/13993003.01193-2022. Print 2023 Mar. PMID 36822634
- See also: Results for CCSJ117X2201 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17681
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=609